CLINICAL TRIAL: NCT03671954
Title: Determining the Effects of Implant Design, Soft Tissue Balance, Neuromuscular Adaptations, and Rehabilitation Strategies on Functional Outcomes and Patient Satisfaction After Total Knee Arthroplasty
Brief Title: Total Knee Arthroplasty Biomechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Orthosensor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201801019; OCR18180 (Other: University of Florida)
Record Dates: First submitted 2018-08-31; First posted 2018-09-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Total Knee Arthroplasty (TKA)
Keywords: knee osteoarthritis; rehabilitation strategies; soft tissue balance
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The intervention group will perform unsupervised home strengthening exercises for the hip abductors in addition to standard physical therapy, while the control group will receive standard physical therapy alone. Subjects will be assigned to one of two groups by block randomization, such that patients receiving each different implant design comprise each block.
Masking Description: Participant, outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TKA Intervention Group (Experimental): The TKA intervention group will perform unsupervised home strengthening exercises for the hip abductors in addition to standard physical therapy.
  Interventions: Behavioral: Home Strengthening Exercises; Other: Standard Physical Therapy
- TKA Control Group (Active Comparator): The TKA control group will receive standard physical therapy alone.
  Interventions: Other: Standard Physical Therapy
- Healthy Control Group (Active Comparator): The Healthy Control Group, aged 49-85 years without any signs of degenerative joint, disease will undergo the preoperative assessments only.
  Interventions: Other: Preoperative Assessments

INTERVENTIONS:
Behavioral: Home Strengthening Exercises — The intervention group will perform unsupervised home strengthening exercises for the hip abductors in addition to standard physical therapy, while the control group will receive standard physical therapy alone.
  Other Names: Hip abductor strengthening program
  Arms: TKA Intervention Group
Other: Standard Physical Therapy — Physician determined standard of care for individual TKA patients.
  Arms: TKA Control Group; TKA Intervention Group
Other: Preoperative Assessments — Assessments will include:
  * TUG (timed up and go test) >12 sec indicates increased fall risk
  * Tandem balance test < 10 sec indicates increased fall risk
  * Sit to Stand test (age based norms)
  * Knee Range Of Motion (ROM)
  * Quadriceps and hamstring strength (MMT or hand held dynamometer)
  * Lower Extremity Functional Score (LEFS questionnaire)
  Arms: Healthy Control Group

SUMMARY:
In total knee arthroplasty (TKA), the relationship between implant design, soft tissue balance, neuromuscular contributions, and rehabilitation strategies on patient satisfaction and functional outcomes is highly complex and poorly understood. The investigators will prospectively study the effects of these factors using in vivo assessments preoperatively, and postoperatively. Computer simulation models will also be used to analyze lower extremity biomechanics.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is the primary treatment for end-stage knee osteoarthritis and effectively relieves pain and improves function after surgery. Nevertheless, as many as 1 in 5 patients are dissatisfied with the postoperative outcome, and knee instability remains one of the top indications for revision surgery. Implant design, soft tissue balance, neuromuscular capabilities, and rehabilitation strategies can all influence postoperative outcomes. However, the relationship between these factors and the most effective therapeutic approach for total knee arthroplasty has yet to be identified. The investigators will study preoperative and postoperative functional measures and patient satisfaction along with implant design and specific intraoperative data, which may help inform a targeted approach for optimal outcomes after total knee arthroplasty and improve future care of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring unilateral TKA for knee osteoarthritis
* No osteoarthritis symptoms in contralateral knee
* Radiographic coronal deformity ≤ 15°
* Preoperative flexion ≥ 90°
* Receiving one of four implants used by UF Orthopaedic surgeons
* Able to walk for a short distance without the use of ambulatory aids
* Healthy Participants:

  1. Age 49-85 years
  2. Healthy with no signs or symptoms of lower limb arthritis or injury
  3. Able to walk for a short distance without the use of ambulatory aids

Exclusion Criteria:

* BMI > 40 kg/m2
* Presence of knee, hip, or ankle prosthesis for either limb
* Presence of hip prosthesis in surgical limb (TKA only subjects)
* History of lower limb or spinal surgery within the last year
* Presence of neurologic or orthopaedic disorders that could affect gait or balance
* Chronic opioid or illicit drug use
* Poorly controlled diabetes (HbA1C > 7 percent)
* Chronic pain syndrome
* Chronic back pain
* Presence of vestibular disorder
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Top declined walking speed before and after TKA. | Tested preoperatively, and once during the two to four months after TKA
  Top walking speed is defined as the maximum speed a patient feels that they can safely walk without running. Patients will walk on an instrumented treadmill declined at seven degrees.
Bilateral isometric quadriceps, hamstrings, and gluteus medius strength before and after TKA | Tested preoperatively, and once during the two to four months after TKA
  Maximum isometric quadriceps, hamstrings, and gluteus medius strength as measured by a dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: MaryBeth Horodyski, EdD, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - UF & Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida
  - UF Health Florida Surgical Center, Gainesville, Florida
  - UF Health at the University of Florida, Gainesville, Florida
  - UF Health Cancer Hospital, Gainesville, Florida